CLINICAL TRIAL: NCT05717530
Title: The Effect of Local Anesthetic Infiltration Into Wound Site or Erector Spina Plan Block on Stress Hormone Response and Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy Surgery
Brief Title: The Effect of Local Anesthetic Infiltration or Erector Spina Plan Block on Stress Hormone Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, murat sahin, principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5234
Record Dates: First submitted 2023-01-24; First posted 2023-02-08 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain; Erector Spinae Plane Block; Inguinal Hernia
Keywords: Cholecystectomy, Laparoscopic; Erector spinae plane block; analgesia; cortisol; prolactin
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- wound site local anesthesic infiltration (Active Comparator): at the end of the operation; 0.5% bupivacaine (1mg/kg) was infiltrated into the fascia muscles and preperitoneal space in equal doses to the wound at the 4 trocar entry site
  Interventions: Procedure: wound site local anesthesic infiltration
- Erector spinae plane block (Active Comparator): : Erector spina block was applied to the group, after the end of the operation, the patients were placed in the left lateral decubitus position and the spinous process of the 8th thoracic vertebra was marked under sterile conditions. After visualizing the spinous process with ultrasound (EsoateMyLab™30 Gold, 8-18 MHz, Genova, Italy), the linear probe (8-12 MHz) was shifted 3 cm laterally from the midline in the cranial-caudal direction. Trapezius, erector spinae muscles, transverse process and pleura were visualized, and 20ml of 0.25% bupivacaine was injected into the validated interval by directing the peripheral nerve block needle in the cranio-caudal direction
  Interventions: Procedure: Erector spina plane block
- Control (No Intervention): There was no intervention.

INTERVENTIONS:
Procedure: wound site local anesthesic infiltration — : at the end of the operation; 0.5% bupivacaine (1mg/kg) was infiltrated into the fascia muscles and preperitoneal space in equal doses to the wound at the 4 trocar entry site.
  Arms: wound site local anesthesic infiltration
Procedure: Erector spina plane block — Erector spina block was applied to the group, after the end of the operation, the patients were placed in the left lateral decubitus position and the spinous process of the 8th thoracic vertebra was marked under sterile conditions. After visualizing the spinous process with ultrasound (EsoateMyLab™30 Gold, 8-18 MHz, Genova, Italy), the linear probe (8-12 MHz) was shifted 3 cm laterally from the midline in the cranial-caudal direction. Trapezius, erector spinae muscles, transverse process and pleura were visualized, and 20ml of 0.25% bupivacaine was injected into the validated interval by directing the peripheral nerve block needle in the cranio-caudal direction.
  Arms: Erector spinae plane block

SUMMARY:
Laparoscopic cholecystectomy is one of the most common operations in abdominal surgery.

Effective analgesia in the postoperative period; It is of great importance in terms of acceleration of recovery, prevention of atelectasis, reduction of endocrine and metabolic stress response, reduction of thromboembolic complications, protection of cognitive functions, prevention of chronic pain development, and reduction of hospital stay . Intravenous paracetamol, NSAID/cyclooxygenase-2 selective inhibitors, opioids, local anesthetic infiltration in the port area, intraperitoneal local anesthetic insufflation or plan blocks can be used in the treatment of postoperative pain after laparoscopic cholecystectomy. Operation, tissue trauma, anesthesia, drugs given to the patient, type of anesthesia, blood loss, temperature changes and pain cause postoperative stress response

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the most common operations in abdominal surgery. Abdominal and shoulder pain are frequently seen in patients in the postoperative period.

Laparoscopic surgery is considered the gold standard in abdominal surgery because of its low cost, less postoperative pain, early mobilization, and short hospital stay. Effective analgesia in the postoperative period; It is of great importance in terms of acceleration of recovery, prevention of atelectasis, reduction of endocrine and metabolic stress response, reduction of thromboembolic complications, protection of cognitive functions, prevention of chronic pain development, and reduction of hospital stay . Intravenous paracetamol, NSAID/cyclooxygenase-2 selective inhibitors, opioids, local anesthetic infiltration in the port area, intraperitoneal local anesthetic insufflation or plan blocks can be used in the treatment of postoperative pain after laparoscopic cholecystectomy. In laparoscopic cholecystectomy operations, the results of pain reduction and analgesic consumption in incisional local anesthetics are variable.

Operation, tissue trauma, anesthesia, drugs given to the patient, type of anesthesia, blood loss, temperature changes and pain cause postoperative stress response .

In various surgeries, regional anesthesia for post-operative purposes, plan blocks, infiltration or insufflation methods were found to suppress the stress response.

In this study, the investigator aimed to compare the effects of local anesthetic infiltration at the wound site and erector spine plane block on stress hormone response and postoperative analgesia in patients who will undergo laparoscopic cholecystectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* who will undergo laparoscopic cholecystectomy
* ASA (American Society of Anesthesiology) I-II
* 18-65 age group
* operated between 08:00-12:00 in the morning

Exclusion Criteria:

* Pregnant,
* Diabetes Mellitus
* Emergency surgery
* ASA (American Society of Anesthesiology)III-IV
* Patients who did not consent to the study,
* History of local anesthetic allergy,
* Coagulation disorder,
* Morbid obesity (body mass index >40 kg/m²),
* Severe organ failure,
* Previous neurological deficit,
* Psychiatric disease,
* Patients with a history of chronic pain
* Who were switched to the open procedure due to surgical complications during the operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Stress hormone response | 5 hour
  Blood was taken and recorded in a yellow capped gel biochemistry tube (SSTTM II Advance Tubes) for the measurement of stress hormone glucose(70-100 mg/dl), prolactin(4.79-23.3µg/dL), and cortisol(60.2-184 µg/dL) 1 hour before and 1 hour after the operation.

SECONDARY OUTCOMES:
Visual Analog Pain Scale | 24 hour
  visual analog for pain consist of a horizontal line, usually 100 mm in length. the left end of the line signifies no pain which is depicted by a smiling face while the right end signifies the worst possible pain with a frowning face. this visual depiction of pain levels helps the patient to communicate about the intensity of their pain.
Analgesia period | 24 hour
  The time from the end of the operation to the first analgesic requirement was determined as the "analgesia period" and this time was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: murat sahin, Principal Investigator — şişli etfal eğitim araştırma hastanesi
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No